CLINICAL TRIAL: NCT02617082
Title: Phase II Study of Partial Breast Irradiation for Low-risk Ductal Carcinoma In Situ After Breast-conserving Surgery
Brief Title: Partial Breast Irradiation for Low-risk Ductal Carcinoma In Situ After Breast-conserving Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoli Yu, professor, Fudan University
Other Study IDs: FDRT-BC004
Record Dates: First submitted 2015-11-21; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; partial breast irradiation; DCIS
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- partial breast irradiation
  Interventions: Radiation: partial breast irradiation

INTERVENTIONS:
Radiation: partial breast irradiation — The prescription dose is 40.5Gy in 15 fractions in 3 weeks.

SUMMARY:
This study is designed to evaluate the feasibility and safety of partial breast irradiation for low risk DCIS after breast-conserving surgery.

DETAILED DESCRIPTION:
Randomized clinical trials have demonstrated that the recurrence of DCIS is low and most of the recurrence occurs around the tumor bed. Besides, cosmetic outcomes are reported better in partial breast irradiation group compared to whole breast irradiation group. However, whether or not partial breast irradiation is safety in DCIS is still unknown. The purpose of this study is to evaluate the feasibility and safety of partial breast irradiation for low risk DCIS after breast-conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18~65 years old
* Pathologically confirmed DCIS, low- or intermediate- grade DCIS: (lesions of ≤2.5 cm diameter, resection margins of at least 3 mm, nuclei grade: 1-2), high grade DCIS: (lesions of ≤1 cm diameter, resection margins of at least 3 mm, nuclei grade: 3)
* Treated with breast conserving surgery
* Tumor bed is labeled with Titanium clips
* No malignancy history
* ECOG score 0~1
* Written informed consent

Exclusion Criteria:

* DCIS of both breast
* invasive breast cancer
* Multicentric disease
* Patients underwent mastectomy
* Previous radiation therapy of breast
* Medical contraindication for radiotherapy
* Pregnant or nursing
* suspicious calcification after surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DCIS breast cancer patients
Sampling Method: Probability Sample
Enrollment: 828 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
ipsilateral breast tumor recurrence | 5 years

SECONDARY OUTCOMES:
occurrence of contralateral breast tumor after PBI | 5 years
Disease free survival | 5 years
Overall survival | 5 years
radiation-induced toxicity of breast assessed by CTCAE v4.0 | baseline, 3 months, 6 months, and every half year to 5 years
Complications | baseline，1，2，3，4，5 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Yu, MD.PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China